CLINICAL TRIAL: NCT00409929
Title: A Randomized, Double-blind, Placebo-controlled, Time Lagged, Parallel Group, Ascending Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral AEB071 Doses Greater Than 500 mg in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of AEB071
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAEB071A2114
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Safety, tolerability, pharmacokinetics, pharmacodynamics, AEB071, healthy subjects, transplantation
MeSH Terms: interventions — sotrastaurin

INTERVENTIONS:
Drug: AEB071

SUMMARY:
This study will evaluate the safety and tolerability of ascending single oral doses greater than 500 mg of AEB071 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects from 18-55 years of age and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram and laboratory tests at screening.
* Female subjects had to either have been surgically sterilized or be postmenopausal.

Exclusion Criteria:

* Smokers
* Use of any prescription drug or over-the-counter medication within 2 weeks prior to dosing, or 2 months for inducers or inhibitors of cytochrome CYP4503A4 (paracetamol acceptable)
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing
* A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome
* History of History of fainting, hypotension when standing up, arrhythmia, acute or chronic bronchospastic disease
* History of clinically significant drug allergy; atopic allergy or a known hypersensitivity to any of the study drugs or drugs similar to the study drugs
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study
* History of immunocompromise (including a positive HIV test result) or drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse or a current positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.

Additional protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ascending single oral doses of AEB071 in healthy subjects.
Maximum Tolerated Dose

SECONDARY OUTCOMES:
Assess the pharmacokinetics of single oral doses of AEB071 at the end of study
Measure inhibition of lymphocytes activation following rising oral doses of AEB071 in healthy subjects after each single dose
Measure the pharmacokinetic/pharmacodynamic relationship of single rising oral doses of AEB071 in healthy subjects after each single dose
Conduct exploratory genomic studies to identify gene expression patterns of blood cells at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Bern, Switzerland